CLINICAL TRIAL: NCT04961788
Title: A Phase 2 Study of Anti-PD1 Antibody Toripalimab Combined With Gemox (Gemcitabine and Oxaliplatin) as First-line Therapy in Patients With Advanced or Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: Anti-PD1 Antibody Toripalimab Combined With Gemox as First-line Therapy in Late-stage Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICC-zs-2021
Record Dates: First submitted 2021-07-07; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic Cholangiocarcinoma; Gemox chemotherapy; PD1 antibody
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemox combined PD1 antibody (Experimental): 1. Toripalimab (240mg) intravenously, the administration time is 60 (+15) minutes, Q3W is administered once.
  2. Gemox chemotherapy D1: oxaliplatin 85mg/m2, gemcitabine 1g/m2 D8: Gemcitabine 1g/m2 Three weeks is a course of treatment, a total of 6-8 courses.
  Interventions: Drug: Gemox combimed PD1 antibody

INTERVENTIONS:
Drug: Gemox combimed PD1 antibody — 1. Toripalimab (240mg) intravenously, the administration time is 60 (+15) minutes, Q3W is administered once.
  2. Gemox chemotherapy D1: oxaliplatin 85mg/m2, gemcitabine 1g/m2 D8: Gemcitabine 1g/m2 Three weeks is a course of treatment, a total of 6-8 courses.

SUMMARY:
To explore the objective response rate and safety of toripalimab combined with Gemox in the first-line treatment of progressive, metastatic or unresectable advanced ICC.

DETAILED DESCRIPTION:
Studies have shown that the Gemox chemotherapy (oxaliplatin + gemcitabine) in patients with advanced biliary tract cancer has an objective response rate (ORR) of 22% (95% CI 6.5-37.4%) and a stable disease rate of 30%. The progression rate was 48%, the tumor progression-free survival (PFS) was 3.9 months and the overall survival (OS) was 7.6 months. In recent years, monoclonal antibodies against programmed cell death protein 1 (PD1) and programmed cell death ligand 1 (PD-L1) such as nivolumab, Pembrolizumab, and Toripalimab. It has shown encouraging effects in the treatment of a variety of solid tumors. For advanced cholangiocarcinoma that cannot be resected or is accompanied by metastasis, NCCN guidelines (NCCN guidelines hepatobiliary cancer, 2020) recommend that the current treatment options are limited, and gemcitabine combined with platinum anti-tumor drugs (cisplatin, oxaliplatin, etc.) are recommended. Chemotherapy regimen as first-line treatment. For those with microsatellite instability, it is recommended to add a PD1 monoclonal antibody. The guidelines also specifically stated that the above recommendations lack evidence support from phase III clinical trials and encourage the development of clinical trial research. PD1 monoclonal antibody combined with chemotherapy in the treatment of advanced ICC may have a better effect than chemotherapy alone. Currently, as a first-line treatment, there is no research report on PD1 monoclonal antibody combined with Gemox in the treatment of advanced ICC.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must sign an informed consent form; 2. Age 18-75 years old, both male and female; 3. ECOG performance status score (PS score) 0 or 1 point; 4. Child-Pugh score A period; 5. Intrahepatic cholangiocarcinoma confirmed by histopathology; agree to provide previously stored tumor tissue specimens or fresh biopsy tumor lesions; 6. Unresectable ICC patients or postoperative diagnosis of ICC recurrence and metastasis, and have not received systemic treatment within 6 months; 7. The functional indicators of important organs meet the following requirements

  1. Neutrophils≥1.5*109/L; platelets≥100*109/L; hemoglobin≥9g/dl; serum albumin≥3g/dl;
  2. Thyroid-stimulating hormone (TSH) ≤ 2 times the upper limit of normal, and T3 and T4 are in the normal range;
  3. Bilirubin ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 3 times the upper limit of normal;
  4. Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 60ml/min (calculated by Cockcroft-Gault formula); 8. The subject has at least 1 measurable lesion (according to RECIST1.1); 9. For women who are not breastfeeding or pregnant, use contraception during treatment or 3 months after the end of treatment.

Exclusion Criteria:

* 1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma, and other malignant components of non-cholangiocarcinoma; 2. Past or simultaneous suffering from other malignant tumors, except for fully treated non-melanoma skin cancer, cervical carcinoma in situ, and thyroid papillary carcinoma; 3. Have used gemcitabine-based chemotherapy or have used PD-1 monoclonal antibody or PD-L1 monoclonal antibody treatment within 6 months; 4. Severe cardiopulmonary and renal dysfunction; 5. Hypertension that is difficult to control with drugs (systolic blood pressure (BP) ≥140 mmHg and/or diastolic blood pressure ≥90mmHg) (based on the average of ≥3 BP readings obtained by ≥2 measurements); 6. Abnormal coagulation function (PT>14s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy; 7. After antiviral treatment, HBV DNA>2000 copies/ml, HCV RNA>1000; 8. A history of esophageal and gastric varices, significant clinically significant bleeding symptoms or a clear tendency to appear within 3 months before enrollment; 9. Active infections requiring systemic treatment; patients with active tuberculosis infection within 1 year before enrollment; a history of active tuberculosis infection more than 1 year before enrollment, and no formal anti-tuberculosis treatment or tuberculosis Still in the active period; 10. Human immunodeficiency virus (HIV, HIV1/2 antibody) positive; 11. A history of psychotropic drug abuse, alcohol or drug abuse; 12. Known to have a history of severe allergies to any monoclonal antibodies, platinum drugs, or gemcitabine; 13. Other factors judged by the investigator may affect the safety of the subjects or the compliance of the trial. Such as serious diseases (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  Objective response rate of advanced and unresectable in intrahepatic cholangiocarcinoma

SECONDARY OUTCOMES:
Safety:The potential side effects | 12 months
  The potential side effects
Overall survival | 18 months
  From the beginning date to the date of death
Progression free survival | 12 months
  From the beginning date to the date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD & PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andre T, Tournigand C, Rosmorduc O, Provent S, Maindrault-Goebel F, Avenin D, Selle F, Paye F, Hannoun L, Houry S, Gayet B, Lotz JP, de Gramont A, Louvet C; GERCOR Group. Gemcitabine combined with oxaliplatin (GEMOX) in advanced biliary tract adenocarcinoma: a GERCOR study. Ann Oncol. 2004 Sep;15(9):1339-43. doi: 10.1093/annonc/mdh351. PMID 15319238
- [Background] Wang FH, Wei XL, Feng J, Li Q, Xu N, Hu XC, Liao W, Jiang Y, Lin XY, Zhang QY, Yuan XL, Huang HX, Chen Y, Dai GH, Shi JH, Shen L, Yang SJ, Shu YQ, Liu YP, Wang W, Wu H, Feng H, Yao S, Xu RH. Efficacy, Safety, and Correlative Biomarkers of Toripalimab in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial (POLARIS-02). J Clin Oncol. 2021 Mar 1;39(7):704-712. doi: 10.1200/JCO.20.02712. Epub 2021 Jan 25. PMID 33492986